CLINICAL TRIAL: NCT05355363
Title: Risk of Metachronous Findings After Detection of Serrated Lesions and High-grade Dysplasia With Surveillance Delay
Acronym: SSL follow-up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22.179
Record Dates: First submitted 2022-04-04; First posted 2022-05-02 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Colon Adenoma
Keywords: sessile serrated polyps; traditional serrated adenomas; high-grade dysplasia; high-risk adenoma; cancer prevention; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: prospective, multi-endoscopist, single center, single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colonoscopy (Experimental): Standard colonoscopy: All optically diagnosed polyps will be removed and sent to the CHUM pathology laboratory for histopathological evaluation according to institutional standards.
  Interventions: Diagnostic Test: Standard Colonoscopy

INTERVENTIONS:
Diagnostic Test: Standard Colonoscopy — Standard colonoscopy: All optically diagnosed polyps will be removed and sent to the CHUM pathology laboratory for histopathological evaluation according to institutional standards.

SUMMARY:
The primary aim of this study is to determine the rate of total metachronous advanced neoplasia (TMAN) detection after index detection of serrated lesions (SL) [sessile serrated polyps (SSPs), traditional serrated adenomas (TSAs)], and metachronous high-risk adenoma (HRA) after index detection of high-grade dysplasia (HGD).

We will use the database of patients diagnosed with SL or HGD at index colonoscopy with a delay in surveillance and determine the risk of advanced lesions (especially high-risk lesion and CRC detection) of these delayed colonoscopies. The aim is to determine the effects of breach of continuity of care in these patients.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) ranks second among worldwide cancer related deaths and third in terms of cancer incidence. Colonoscopy-based screening programs have been established to reduce CRC morbidity and mortality. Multiple guidelines have established surveillance recommendations for repeat colonoscopies based on findings at index colonoscopy. Serrated lesions (SLs), including sessile serrated polyps/adenomas (SSP) and traditional serrated adenomas (TSA) have become of increased interest for their role as precursors of CRC. The optimal timing of follow-up colonoscopies after detection of SLs has been controversial as studies looking into optimal surveillance timing are lacking. The US Multi Society Task Force (USMSTF) 2020 guidelines recommend 5-10y surveillance intervals for detection of 1-2 SSPs, 3-5y for 3-4 SSPs, 3y for >4 SSPs or TSA. In contrast, the 2020 European Society of Gastrointestinal Endoscopy (ESGE) Guidelines state that 1-10mm SLs do not require follow-up. It is unclear what the appropriate surveillance intervals is for patients with SLs which is evidenced by diverging recommendations from USMSTF/ESGE. High-grade dysplasia (HGD) is an exceedingly rare finding in colorectal polyps. The current literature on the yield of colonoscopy after index HGD is sparse, with conflicting data on risk of metachronous HRA due to low numbers of included HGD leading to high variability in reported outcomes.

Patient with SL or HGD diagnosed from 2010-2022 will be gathered from the pathology department to determine which patients lack follow-up during these years. Patients with lack of follow-up will be contacted by phone, then invited to undergo follow-up colonoscopy as part of our routine clinical follow-up of these patients' files.

In addition to the primary and secondary endpoints, data collected will include patient age; sex; ASA class; past medical history; family history of CRC; procedure date; name of endoscopist; colonoscopy indication; BBPS score; withdrawal time; adenoma and polyp detection rate at index and follow-up colonoscopy; completeness of polypectomy; polyp location, size, surface, morphology (Paris classification), histopathology; complications, immediate and late (14 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients 45-80 who underwent colonoscopy from 2009 to 2022 at the Montreal University Hospital Center (CHUM) with 1+ SL or HGD detected at index colonoscopy and lacking follow-up within or beyond the surveillance interval recommended by 2020 USMSTF guidelines.

Exclusion Criteria:

* 1) Patients with a diagnosis of inflammatory bowel disease;
* 2) Hereditary CRC syndromes;
* 3) CRC at index colonoscopy;
* 4) Serrated polyposis syndrome;
* 5) Life expectancy too short to benefit from colonoscopy;
* 6) Follow-up colonoscopy not yet due according to USMSTF guidelines. Patients with concomitant HRA and SL at index will be invited to participate if the index (or last) colonoscopy was performed more than 1 year ago. This is based on the high rates of HRA we identified in our retrospective study posing increased risks for these patients.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of TMAN detection after index detection of serrated lesions | 1 year
  the rate of total metachronous advanced neoplasia (TMAN) detection after index detection of serrated lesions [sessile serrated polyps (SSPs), traditional serrated adenomas (TSAs)]
Rate of metachronous high-risk adenoma (HRA) after index detection of high-grade dysplasia (HGD) | 1 year
  the rate of metachronous high-risk adenoma (HRA) after index detection of high-grade dysplasia (HGD)

SECONDARY OUTCOMES:
Rate of T-MAN detection for concomitant index SSP+low-risk adenoma (LRA); index SSP+ high-risk adenoma (HRA); index SSP alone | 1 year
  The rate of T-MAN detection for concomitant index SSP+low-risk adenoma (LRA); index SSP+ high-risk adenoma (HRA); index SSP alone
Rate of T-MAN detection according to number, size, location, and dysplasia status of index SSPs | 1 year
  The rate of T-MAN detection according to number, size, location, and dysplasia status of index SSPs
Rate of metachronous HRA detection for index HGD alone | 1 year
  The rate of metachronous HRA detection for index HGD alone
Rate of metachronous HRA detection for index HGD according to number, size, location, of index HGD | 1 year
  The rate of metachronous HRA detection for index HGD according to number, size, location, of index HGD
Rate of metachronous high-risk serrated lesion (SL) for concomitant index SSP+LRA; index SSP+HRA; index SSP alone; index SSP all synchronous findings included; index TSA a ll synchronous findings included | 1 year
  The rate of metachronous high-risk serrated lesion (SL) for concomitant index SSP+LRA; index SSP+HRA; index SSP alone; index SSP all synchronous findings included; index TSA all synchronous findings included
Rate of metachronous high-risk SL detection according to number, size, location, and dysplasia status of index SSPs | 1 year
  The rate of metachronous high-risk SL detection according to number, size, location, and dysplasia status of index SSPs
Rate of metachronous HRA for concomitant index SSP+LRA; index SSP+HRA; index SSP alone; index SSP all synchronous findings included; index TSA all synchronous findings included | 1 year
  The rate of metachronous HRA for concomitant index SSP+LRA; index SSP+HRA; index SSP alone; index SSP all synchronous findings included; index TSA all synchronous findings included
Rate of metachronous HRA detection according to number, size, location, and dysplasia status of index SSPs | 1 year
  The rate of metachronous HRA detection according to number, size, location, and dysplasia status of index SSPs
Rate of T-MAN and metachronous HRA detection for the serrated lesion (SL) and HGD groups | 1 year
  The rate of T-MAN and metachronous HRA detection for the serrated lesion (SL) and HGD groups stratified by number of years of surveillance delay
Rate of metachronous advanced SL and metachronous HRA detection for the serrated lesion (SL) group | 1 year
  The rate of metachronous advanced SL and metachronous HRA detection for the serrated lesion (SL) group stratified by number of years of delay at time of endoscopy from surveillance intervals recommended by guidelines
Adenoma detection rates (ADR) and advanced adenoma detection rates at follow-up | 1 year
  Adenoma detection rates (ADR) and advanced adenoma detection rates at follow-up stratified by number of years of delay at time of endoscopy from surveillance intervals recommended by guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, Md, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No